CLINICAL TRIAL: NCT01937494
Title: Are Technicians Showing Bronchial Hyperreactivity Able to Safely Perform Bronchial Provocation Tests?
Brief Title: Bronchial Hyperreactivity During Histamine Passive Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, CCA, pneumologie, Centre Hospitalier Universitaire Saint Pierre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AK/13-03-34/4235
Record Dates: First submitted 2013-08-29; First posted 2013-09-09 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Asthma; Bronchial Hyperresponsiveness
Keywords: asthma; bronchial hyperresponsiveness; histamine challenge test; spirometry
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- asthma patients (Experimental): patients who show a positive response at the first dos of histamine challenge test will be enrolled
  Interventions: Drug: histamine-benzylic alcohol (magistral preparation)

INTERVENTIONS:
Drug: histamine-benzylic alcohol (magistral preparation) — passive exposure to histamine during a bronchial hyperresponsiveness challenge

SUMMARY:
Bronchial hyperresponsiveness consists in excessive response to bronchial stimuli.Bronchial challenge test is used to confirm/exclude asthma (metacholine or histamine).Protection are used to avoid passive exposure of the technicians performing the test, despite the absence of evidence that they could develop a bronchoconstriction even if they suffer from BHR.The purpose of the study is to determine if patients with a high level of bronchial hyperreactivity and exposed passively to histamine during a bronchial challenge, are developing a bronchoconstriction, when placed in the same conditions that the technicians performing these tests.

DETAILED DESCRIPTION:
Bronchial hyperresponsiveness (BHR) consists in excessive response to bronchial stimuli.Bronchial challenge test is used to confirm/exclude asthma.BHR is also present in other diseases such as allergic rhinitis, Chronic Obstructive pulmonary disease,heart failure..

Thes test is performed with metacholine or histamine with spirometric documented response to incremental doses.Protection are used to avoid passive exposure of the technicians performing the test, despite the absence of evidence that they could develop a bronchoconstriction if they suffer from BHR.

The purpose of the study is to determine if patients, newly diagnosed with a high level of bronchial hyperreactivity and exposed passively to histamine during a bronchial challenge, are reacting to histamine when placed in the same conditions that the technicians performing these tests.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with positive histamine challenge test (first dose)

Exclusion Criteria:

* other active respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
spirometric values in patients exposed passively to histamine during BHR challenge | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Principal Investigator — CHU ST Pierre
Locations (1):
- service de pneumologie, CHU St Pierre, Brussels, Belgium